CLINICAL TRIAL: NCT07027449
Title: Implementing Pathways to Identify and Address Employment Concerns Among People With Cancer Across Diverse Clinical Settings
Brief Title: Connecting People With Cancer to Employment Support
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00161657
Record Dates: First submitted 2025-05-27; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Cancer
Keywords: employment; social needs; screening
MeSH Terms: conditions — Neoplasms | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening and Referral Workflow (Experimental)
  Interventions: Behavioral: Screening and Referral Workflow

INTERVENTIONS:
Behavioral: Screening and Referral Workflow — The Screening and Referral Workflow intervention will include screening eligible patients for employment-related needs and referring those who require support to community-based employment resources.

SUMMARY:
The goal of this clinical trial is to learn if a clinical workflow that screens adult patients with cancer for challenges at work and refers them to supportive resources is feasible, appropriate, and acceptable to patients and staff members in 2 cancer care settings. The main questions it aims to answer are:

Is the clinical workflow feasible and acceptable to participants? Are study procedures feasible and acceptable to participants?

Patient participants will complete 2 surveys: 1 at the time of enrollment and 1 six months later.

DETAILED DESCRIPTION:
Investigators will conduct a prospective single-arm study at 2 sites to pilot and iteratively adapt a clinical workflow intervention, implementation strategies, and associated study procedures. Investigators will implement the clinical workflow intervention across each study site, then recruit consecutive patients (n=50) to complete patient-reported measures at 2 time points (T1: enrollment; T2: 6-month follow-up. Investigators will recruit staff members (n=20) to complete survey measures at 2 time points (T1: beginning of pilot study period; T2: end of pilot study period).

ELIGIBILITY:
Eligible Patients:

* visiting a participating medical or radiation oncology clinic for new diagnosis, treatment, or follow-up of any type of cancer;
* employed at the time of cancer diagnosis;
* age 18 or older;
* able to give full informed consent;
* able to communicate in English or Spanish.

Eligible Staff:

* age 18 or older;
* employed at one of the participating clinical sites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2028-01 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Enrollment Rate | Baseline
  T1 survey enrollment rate among eligible patients and staff
Follow-up Survey Completion Rate | 6 months
  Rate of study survey completion within 18 days of the 6-month follow-up timepoint
Staff-reported Feasibility of Intervention | Approximately 9 months
  Proportion of staff disagreeing with one or more Feasibility of Intervention Measure items
Acceptability of Intervention: Staff | Approximately 9 months
  Proportion of staff disagreeing with one or more Acceptability of Intervention Measure items
Acceptability of Intervention: Patients | Baseline; 6 months
  Proportion of patients providing negative ratings for one or more Theoretical Framework of Acceptability questionnaire items
Employment Concerns Screening | Baseline
  Proportion of eligible patients screened for employment concerns

SECONDARY OUTCOMES:
Employment status | Baseline; 6 months
  Patient-reported employment status using the US Census Bureau's American Community Survey employment status items
Sick leave duration | Baseline; 6 months
  Patient-reported sick leave duration reported in days
Health-related quality of life | Baseline; 6 months
  Patient-reported quality of life using the EQ-5D-5L scale. Scores range 1-5, with higher scores indicating poorer quality of life (worse outcome).
Health insurance status | Baseline; 6 months
  Patient-reported health insurance status using the US Census Bureau's American Community Survey health insurance status items
Self-efficacy | Baseline; 6 months
  Patient-reported self-efficacy using the General Self-Efficacy Scale. Scores range 10-40, with higher scores indicating more self-efficacy (better outcome).
Financial toxicity | Baseline; 6 months
  Patient-reported financial toxicity using the COST measure. Scores range 0-48, with higher scores indicating more financial toxicity (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Rachel C. Forcino, PhD, MSc, Principal Investigator — University of Kansas Medical Center

IPD SHARING:
Plan to Share IPD: No